CLINICAL TRIAL: NCT02703883
Title: Effects of Body Weight-supported Treadmill Training on Center of Mass Control in Spinal Cord Injury, Measured With Inertial Sensors
Brief Title: Body Weight Support in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Torres, MSc, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLC-1
Record Dates: First submitted 2016-02-29; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Body Weight Support (Experimental): Treatment protocol consisted of 18 training sessions on the BWST, three times a week, every session included three sets of six minutes of locomotion with rest intervals of 2 min of rest.
  Interventions: Device: BWST

INTERVENTIONS:
Device: BWST — BWST (six weeks, 3 times/week)

SUMMARY:
The purpose of this study was to evaluate the effectiveness of body weight-supported treadmill (BWST) training on static balance impairment in adults with incomplete spinal cord injury (SCI) in chronic stage

DETAILED DESCRIPTION:
The individuals who participated in this study were subjects with SCI with more than twelve months of evolution. All were classified as incomplete injury class C or D according to the American Spinal Injury Association (ASIA). Each received training on a BWST for six weeks. Two measures of stance balance were performed during the training protocol. The first measure was made before entering the training protocol; the final measure was implemented once the gait training on BWST protocol was completed. For instrumented stance balance testing, small wireless inertial motion sensors (OPAL sensors, APDM Inc., Portland, OR) were placed on the subjects' waist. Subjects performed instrumented stance with their eyes opened (iSway). Outcome measures were recorded and automatically generated using Mobility Lab software (APDM Inc., Portland, OR). Measures included the root mean square of sway and jerk (normalized to the range of acceleration amplitude).

ELIGIBILITY:
Inclusion Criteria:

* SCI with more than twelve months of evolution.
* ASIA C and D

Exclusion Criteria:

* Patients with tracheostomy
* Patients with severe respiratory, cognitive and cardiovascular comorbidities
* Patients with peripheral nerve injury in lower limbs
* Patients with traumatic head injury

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Jerk (Derivative of the acceleration of the mass center as marker oscillation of the control the center of mass) | 6 weeks
  The jerk is measure with a instrumented stance testing. For this test, we use small wireless inertial sensors (OPAL sensor, APDM, Inc. Portland, OR). This outcome is recorded automatically generated using Mobility Lab Software (APDM Inc., Portland, OR).

SECONDARY OUTCOMES:
Walking Index for Spinal Cord Injury (WISCI) scale | 6 weeks
  The WISCI is a walking scale, that measures the independence of walking based on the use of devices.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Covarrubias, Principal Investigator — Clinica Los Coihues
Locations (1):
- Clínica Los Coihues, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Covarrubias-Escudero F, Rivera-Lillo G, Torres-Castro R, Varas-Diaz G. Effects of body weight-support treadmill training on postural sway and gait independence in patients with chronic spinal cord injury. J Spinal Cord Med. 2019 Jan;42(1):57-64. doi: 10.1080/10790268.2017.1389676. Epub 2017 Oct 23. PMID 29058553